CLINICAL TRIAL: NCT04649996
Title: Variation of Incidence and Clinical Presentation of Acute Appendicitis During a Pandemic.
Brief Title: Variation in Acute Appendicitis During COVID-19 Pandemic in Italy
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: Appendicitis-pandemic
Record Dates: First submitted 2020-12-01; First posted 2020-12-02 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy; Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pandemic period: patients admitted in hospital for acute appendicitis
  Interventions: Procedure: Appendectomy
- control period: patients admitted in hospital for acute appendicitis
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — comparison between operative and conservative treatment
  Other Names: Conservative treatment

SUMMARY:
retrospective observational study of variation in incidence and clinical presentation of appendicitis during the pandemic in northern Italy, compared with the same period in the previous 2 years.

ELIGIBILITY:
Inclusion Criteria:

* acute appendicitis

Exclusion Criteria:

* other diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted in hospital for acute appendicitis
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
complicated appendicitis | 2 months
  Number of patients with complicated acute appendicitis

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Policlinico San Pietro, Ponte San Pietro, BG
  - Ospedale Manzoni, Lecco, LC
  - ASST Monza, Monza, MB
  - Ospedale San Raffaele, Milan, Mi
  - ASST Lodi, Lodi
  - Azienda ospedaliero-universitaria Pisana,Ospedale Cisanello, Pisa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ceresoli M, Coccolini F, Magnone S, Lucianetti A, Bisagni P, Armao T, Ansaloni L, Zago M, Chiarugi M, Catena F, Braga M; Appendicitis-COVID study group. The decrease of non-complicated acute appendicitis and the negative appendectomy rate during pandemic. Eur J Trauma Emerg Surg. 2021 Oct;47(5):1359-1365. doi: 10.1007/s00068-021-01663-7. Epub 2021 Apr 12. PMID 33844036